CLINICAL TRIAL: NCT05873088
Title: Effects of Isometric Versus Isotonic Exercise in Female Patients With Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/538
Record Dates: First submitted 2023-03-18; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric (Other)
  Interventions: Diagnostic Test: Isometric
- Isotonic Exercise (Experimental)
  Interventions: Diagnostic Test: Isotonic Exercise

INTERVENTIONS:
Diagnostic Test: Isometric — Effects of Isometric Exercise in Female Patients With Osteoarthritis
  Arms: Isometric
Diagnostic Test: Isotonic Exercise — Effects of Isotonic Exercise in Female Patients With Osteoarthritis
  Arms: Isotonic Exercise

SUMMARY:
to find out the Effects of Isometric Versus Isotonic Exercise in Female Patients With Osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Female patients with osteoarthritis Age group of 35 to 60

Exclusion Criteria:

* Patients admitted in ICU or HDU Patients with any mental illness

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC Scale | 6 Months
  Isometric Versus Isotonic Exercise in Female Patients With Osteoarthritis by using WOMAC Scale
VAS score | 6 Months
  Isometric Versus Isotonic Exercise in Female Patients With Osteoarthritis by using VAS score

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudhary Muhammad Akram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No